CLINICAL TRIAL: NCT02602509
Title: Evaluating Celecoxib Activity in Mycobacterium Tuberculosis: A Whole Blood Bactericidal Activity Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Celecoxib_WBA
Record Dates: First submitted 2015-11-06; First posted 2015-11-11 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2015-11

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Celecoxib; Rifampin; Pyrazinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Celecoxib plus rifampicin group (Experimental): Visit 1: Celecoxib 400mg Visit 2: Rifampicin 10mg/kg Visit 3: Celecoxib 400mg PLUS rifampicin 10mg/kg
  Interventions: Drug: Celecoxib; Drug: Rifampicin
- Celecoxib plus pyrazinamide group (Experimental): Visit 1: Celecoxib 400mg Visit 2: Pyrazinamide 25mg/kg Visit 3: Celecoxib 400mg PLUS pyrazinamide 25mg/kg
  Interventions: Drug: Celecoxib; Drug: Pyrazinamide

INTERVENTIONS:
Drug: Celecoxib
  Other Names: Celebrex
Drug: Rifampicin
  Other Names: Rifampin
  Arms: Celecoxib plus rifampicin group
Drug: Pyrazinamide
  Arms: Celecoxib plus pyrazinamide group

SUMMARY:
The purpose of this study is to evaluate the bactericidal activity against Mycobacterium tuberculosis of celecoxib in combination with established drugs used to treat tuberculosis (TB). Pharmacokinetics (PK) and whole blood bactericidal activity (WBA) will be measured in healthy volunteers following administration of the study drugs alone and in combination.

DETAILED DESCRIPTION:
The whole blood bactericidal activity (WBA) assay is an ex vivo model for measuring the combined effects of administered drugs, host factors and strain factors on mycobacterial sterilisation. If performed in parallel with PK measurements, the method can be used to evaluate the effect of drugs throughout the dosing cycle. Celecoxib is a COX-2 inhibitor with immuno-modulatory properties important in the host defence against tuberculosis (TB). The aim of this trial is to investigate the effect on WBA of manipulation of the host response to TB using celecoxib, in combination with established TB drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 21 years and below 60 years old
2. Male or female willing to comply with the study visits and procedures
3. Willing and able to provide written informed consent

Exclusion Criteria:

1. Women who are currently pregnant or breastfeeding
2. Body weight below 50kg
3. Clinical signs of active TB in the opinion of the investigator
4. Previous hypersensitivity, intolerance or allergy to rifampicin, pyrazinamide, COX-2 inhibitors, non-steroidal anti-inflammatory drugs or sulfonamides
5. Current use of any drugs or medication known to have an interaction with rifampicin, pyrazinamide or celecoxib
6. Current use or use in the last 2 weeks of non-steroidal anti-inflammatory drugs or COX-2 inhibitors
7. Current use or use in the last 2 weeks of any drugs, over the counter or herbal preparations that are known or potential inhibitors or inducers of cytochrome P450 enzymes
8. Evidence of renal or hepatic dysfunction or any clinically significant deviation from normal during screening including laboratory determinations
9. Known hepatic disease, recent hepatitis (within last 6 months) or alcohol abuse
10. Known cardiovascular disease, heart failure, stroke or current cardiovascular risk factors
11. Known peptic ulcer disease, previous gastrointestinal bleed or current risk factors for gastrointestinal events
12. Acute or previous gout, acute porphyria
13. Any other significant condition that would, in the opinion of the investigator, compromise the volunteer's safety or outcome in the trial
14. Current participation in other clinical intervention trial or research protocol

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Log change CFU.day (cumulative over 8 hours) calculated from Mycobacteria Growth Indicator Tube (MGIT) Time to Positivity | 8 hours
  Cumulative whole blood bactericidal activity (WBA)

SECONDARY OUTCOMES:
Plasma concentrations of study drugs to determine the Area Under the Curve (AUC) | 8 hours
Plasma concentrations of study drugs to determine the Maximum Plasma Concentration (Cmax) | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Paton, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore